CLINICAL TRIAL: NCT05395338
Title: 1-year Clinical Outcomes After Intravenous Rt-PA for Chinese AIS Patients
Brief Title: 1-year Clinical Outcomes in Recombinant Tissue Plasminogen Activator (Rt-PA) Treated Chinese Acute Ischaemic Stroke (AIS) Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 0135-0350
Record Dates: First submitted 2022-05-25; First posted 2022-05-27 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IV rt-PA cohort: Patients who received IV rt-PA within 4.5 hours of symptom onset
  Interventions: Drug: rt-PA
- Non-reperfusion cohort: Patients who arrived or were admitted to the hospital within4.5 hours of symptom onset and did not receive any reperfusion treatment

INTERVENTIONS:
Drug: rt-PA — Recombinant Tissue Plasminogen Activator
  Groups: IV rt-PA cohort

SUMMARY:
The objective of the study is to find out the 1-year clinical outcomes among Acute Ischaemic Stroke (AIS) patients who were treated with intravenous (IV) Recombinant Tissue Plasminogen Activator (rt-PA) within 4.5 hours of symptom onset compared with those who arrived or were admitted to the hospital within 4.5 hours of symptom onset and did not receive any reperfusion treatment in a real-world clinical setting.

ELIGIBILITY:
Inclusion criteria:

* Patients registered in the ZSQCC platform from Jan 2017 to Mar 2020
* ≥ 18 years of age
* Diagnosed with AIS at admission
* Arrived or admitted to the hospital within 4.5 hours of symptom onset
* If treated with IV rt-PA: received IV rt-PA within 4.5 hours of symptom onset

Exclusion criteria:

* Documented Intravenous Thrombolysis (IVT) contraindication except age to IV rt-PA treatment according to the Summary of Product Characteristics (SmPC)
* Missing any one of the key data (age, gender, baseline National Institutes of Health Stroke Scale [NIHSS], time of symptom onset, time of hospital arrival or admission, IVT or not, time of IV rt-PA treatment)
* Received thrombolysis agents other than rt-PA (urokinase, tenecteplase, recombinant plasminogen activator, prourokinase, streptokinase)
* Received endovascular treatment
* Received IV rt-PA after 4.5 hours of symptom onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, AIS patient data from 80 stroke centres in the Zhejiang Stroke Quality Control Centre (ZSQCC) platform from January 2017 to March 2020 will be used.
Sampling Method: Non-Probability Sample
Enrollment: 12551 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boehringer Ingelheim (China) Investment Co., ltd., Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-interventional study (NIS) based on existing data collected from the Zhejiang Stroke Quality Control Centre (ZSQCC) platform of Acute Ischaemic Stroke (AIS) patients aged ≥18 years in China aimed to compare the 1-year mortality of AIS patients treated with intravenous (IV) Recombinant Tissue Plasminogen Activator (rt-PA) within 4.5 hours of symptom onset versus those who arrived or were admitted to the hospital within 4.5 hours of symptom onset and did not receive reperfusion treatment.
Pre-assignment Details: Between January 2017 and March 2020, 98,330 AIS patients were registered in the ZSQCC platform. A total of 12,551 patients were included in the study, with 6,494 of them matched 1:1 (3,247 in the IV Rt-PA Cohort and 3,247 in the Non-reperfusion Cohort) based on baseline characteristics using the propensity score matching (PSM) method. Only the propensity score-matched patients as described here were used for the data analyses.
Groups:
- Non-reperfusion Cohort: Patients who arrived or were admitted to the hospital within 4.5 hours of symptom onset and did not receive any reperfusion treatment
Period: Overall Study
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort
Started | 8014 | 4537
Propensity Score Matched Patients | 3247 | 3247
Completed | 8014 | 4537
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Propensity score matched (PSM) cohorts of AIS patients between the IV rt-PA and non-reperfusion groups (1:1). Patients >= 18 years old and registered in the Zhejiang Stroke Quality Control Centre (ZSQCC) platform from Jan 2017 to Mar 2020.
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort | Total
Number analyzed (Participants) | 3247 | 3247 | 6494
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.2 (11.6) | 70.2 (12.9) | 70.2 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1303 | 1318 | 2621
  Male | 1944 | 1929 | 3873
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Race and Ethnicity were not collected from any participant. Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality at 1 Year (Percentage of Patients With Modified Rankin Scale (mRS) Score =6)
Description: The modified Rankin Scale (mRS) is used for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
  The scale runs from 0-6, from 'perfect health without symptoms' to 'death'. 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Time Frame: Up to 1 year.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort
Number analyzed (Participants) | 3247 | 3247
Percentage of Participants | 11.1 [10.0 to 12.2] | 12.2 [11.1 to 13.3]
Statistical Analysis 1: Comparison: IV Rt-PA Cohort vs Non-reperfusion Cohort; Test type: Other — cox proportional hazards models with stratification by matching pairs; p = 0.183, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.78 to 1.05] — rt-PA/non reperfusion

2. Secondary Outcome: Percentage of Patients With Functional Independence (mRS Score 0 to 2) at 1 Year
Description: as for outcome 1
Time Frame: Up to 1 year.
Population: Propensity score matched (PSM) cohorts of AIS patients between the IV rt-PA and non-reperfusion groups (1:1). Patients >= 18 years old and registered in the ZSQCC platform from Jan 2017 to Mar 2020. Only patients with available mRS data for this outcome were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort
Number analyzed (Participants) | 3083 | 3083
Percentage of Participants | 70.9 [69.3 to 72.5] | 66.4 [64.7 to 68.0]
Statistical Analysis 1: Comparison: IV Rt-PA Cohort vs Non-reperfusion Cohort; Test type: Other — Conditional logistic regression models with stratification by matching pairs; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [1.12 to 1.39]

3. Secondary Outcome: Percentage of Patients With Favourable Outcome (mRS Score 0 to 1) at 1 Year
Description: as for outcome 1
Time Frame: Up to 1 year.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort
Number analyzed (Participants) | 3083 | 3083
Percentage of participants | 59.5 [57.8 to 61.2] | 54.6 [52.8 to 56.3]
Statistical Analysis 1: Comparison: IV Rt-PA Cohort vs Non-reperfusion Cohort; Test type: Other — Conditional logistic regression models with stratification by matching pairs; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [1.11 to 1.36] — rt-PA/non reperfusion

4. Secondary Outcome: Percentage of Patients With mRS Score 5 to 6 at 1 Year
Description: as for outcome 1
Time Frame: Up to 1 year.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort
Number analyzed (Participants) | 3083 | 3083
Percentage of participants | 15.9 [14.6 to 17.2] | 20.3 [18.9 to 21.7]
Statistical Analysis 1: Comparison: IV Rt-PA Cohort vs Non-reperfusion Cohort; Test type: Other — Conditional logistic regression models with stratification by matching pairs; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.64 to 0.83] — rt-PA/non reperfusion

5. Secondary Outcome: Distribution of mRS Score at 1 Year
Description: The modified Rankin Scale (mRS) is used for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Clinicians give the mRS score per the clinical diagnosis/symptom to the patient. There is no calculation for this endpoint or each individual components.
  The scale runs from 0-6, from 'perfect health without symptoms' to 'death'.
Time Frame: Up to 1 year.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort
Number analyzed (Participants) | 3083 | 3083
Score on a scale | 1.8 (2.0) | 2.0 (2.1)
Statistical Analysis 1: Comparison: IV Rt-PA Cohort vs Non-reperfusion Cohort; Test type: Other — Ordinal logistic regression models; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.77 to 0.93] — rt-PA/non reperfusion

ADVERSE EVENTS:
Time Frame: All-Cause-mortality: From the patient registration in the ZSQCC platform (between January 2017 and March 2020) to 1-year follow-up, up to 1 year.
Description: This is a non-interventional study (NIS) based on existing data from the Zhejiang Stroke Quality Control Centre (ZSQCC) platform. No adverse events were collected on an individual case level. Serious Adverse Events and Other Adverse Events are not collected in the database. "0" total Number of Participants at Risk means "Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed".
  All-Cause Mortality is an outcome of this study and thus additionally reported below.
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort
All-Cause Mortality (participants affected / at risk) | 360/3247 | 396/3247
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This was a non-interventional study (NIS) based on existing data, although Propensity Score Matching (PSM) was used, we cannot rule out the influence of other unmeasured confounding factors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT05395338/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT05395338/SAP_001.pdf